CLINICAL TRIAL: NCT05086458
Title: Impact of Probiotics Supplement on the Gut Microbiota in Caesarean-born Infants: an Open-label Single-center Randomized Parallel Controlled Study
Brief Title: Impact of Probiotics Supplement on the Gut Microbiota in Caesarean-born Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Director, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHSYEK-001
Record Dates: First submitted 2021-08-18; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Gut Microbiota
Keywords: gut microbiota; probiotics; infant; cesarean section
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention): the patients in this arm will not receive probiotics.
- Dietary Supplement (Experimental): the patients in this arm will receive probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus, Enterococcus faecalis for 2 weeks.
  Interventions: Dietary Supplement: probiotics

INTERVENTIONS:
Dietary Supplement: probiotics — probiotics blend of Bifidobacterium longum, Lactobacillus acidophilus, Enterococcus faecalis
  Arms: Dietary Supplement

SUMMARY:
The purpose of this study is to evaluate the effect of probiotics on the gut microbiota of infants born by cesarean section.

DETAILED DESCRIPTION:
This study aims to examine the impact of probiotics administration on the gut microbiota of infants born by cesarean section. Birth,14 days and 42 days data will be collected and put into analysis to provide some suggestions on the probiotics use in the clinical for the infants born by cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born by caesarean section

Exclusion Criteria:

* Gestational weeks <37 Birth weight <2500g or ≥4000g History of asphyxia anoxia at birth With congenital metabolic diseases or hereditary diseases With gastrointestinal diseases With infectious diseases

Ages: 1 Hour to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-10-17 (Estimated); Study Completion 2021-10-17 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiota at 42 days between no intervention group and experimental group. | 42 days
  Study the microbiota change of stool samples at 42 days between no intervention group and experimental group.
Change in gut microbiota at 14 days between no intervention and experimental group. | 14 days
  Study the microbiota change of stool samples 14 days between no intervention group and experimental group.

SECONDARY OUTCOMES:
Change in gut microbiota at birth between no intervention and experimental group. | birth
  Study the microbiota change of stool samples at birth between no intervention group and experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Huanlong Qin, MD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Rong Yang, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gong Y, Zhong H, Wang J, Wang X, Huang L, Zou Y, Qin H, Yang R. Effect of Probiotic Supplementation on the Gut Microbiota Composition of Infants Delivered by Cesarean Section: An Exploratory, Randomized, Open-label, Parallel-controlled Trial. Curr Microbiol. 2023 Sep 15;80(11):341. doi: 10.1007/s00284-023-03444-4. PMID 37712964